CLINICAL TRIAL: NCT06889948
Title: Daratumumab in Monoclonal Gammopathy of Renal Significance in Finland
Brief Title: The Effect of Daratumumab in Patients with Monoclonal Gammopathy of Renal Significance (MGRS) in Finland
Acronym: DAMOCLES
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Janssen, L.P. - Investigator Initiated Studies Program (Unknown)
Responsible Party: Principal Investigator, Minna Seppälä, MD, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20221; 2021-005856-12 (EudraCT Number)
Record Dates: First submitted 2025-02-14; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Kidney Failure; Paraproteinemias; Glomerulonephritis
Keywords: Monoclonal gammopathy of renal significance; daratumumab
MeSH Terms: conditions — Renal Insufficiency; Paraproteinemias; Glomerulonephritis | interventions — daratumumab

STUDY DESIGN:
Intervention Model Description: All patients will receive either fixed-dose daratumumab as a single agent therapy or fixed-dose daratumumab combined with stem cell transplantation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daratumumab as a single agent therapy (Active Comparator): Daratumumab
  Interventions: Drug: Daratumumab
- Daratumumab combined with stem cell transplantation (Active Comparator): Daratumumab in combination with stem cell transplantation
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — All patients will receive either fixed-dose daratumumab as a single agent therapy or fixed-dose daratumumab combined with stem cell transplantation.

SUMMARY:
The goal of this clinical trial is to learn if drug daratumumab works to treat kidney diseases other than AL-amyloidosis that fall under the category of monoclonal gammopathy of renal significance (MGRS).

The main questions it aims to answer are:

Does daratumumab have an effect on the patients' renal function or the amount of proteinuria?

Does daratumumab have an effect on the hematological endpoints evaluated by minimal residual disease (MRD) and the difference between involved and uninvolved free light chain (dFLC)?

Also changes in quality of life (according to EORTC QLQ-C30) and mechanism of complement system activation are evaluated. The number of patiets with partial or very good partial hematological remission and the number of patients with adverse events related to daratumumab are also recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 18 years of age
2. Subject has provided informed consent prior to initiation of the study or subject's legally acceptable representative has provided informed consent prior to the study when the subject has any kind of condition that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent.
3. Renal biopsy confirmed MGRS-disease

   * Renal biopsy must not be older than 3 months before informed consent. However, if renal biopsy is older than 3 mo and the study team is convinced that major histological changes have not occurred, a biopsy older than that can exceptionally be accepted.
   * Renal transplant patients are allowed
4. Amount of proteinuria ≥ 500 mg/24 h OR eGFR ≥ 20 ml/min prior to the study
5. Previous anticlonal treatment is allowed if deemed ineffective

Exclusion Criteria:

1. Myeloma or systemic AL amyloidosis (smoldering myeloma sized plasma cell clone is allowed when in association with a documented MGRS condition and AHL amyloidosis and AH amyloidosis are included)
2. Cancer that requires treatment,
3. MGRS related to B-cell malignant disorders,
4. Known HIV infection, active hepatitis C infection (subjects with hepatitis C that achieve a sustained virologic response after antiviral therapy are allowed), or hepatitis B infection (subjects with hepatitis B surface antigen or core antibody that achieve sustained virologic response (PCR negativity in HBVNh) with antiviral therapy are permitted with a requirement for regular monitoring for reactivation for the duration of treatment on the study),
5. Pregnancy or breastfeeding,
6. Cyclophosphamide within 6 months of enrollment, or oral high-dose prednisone or equivalent within 6 weeks of enrollment;

   * prednisone or its equivalent at a dosage of ≤10 mg daily for a condition unrelated to MGRS (e.g. asthma or gout) allowed.
   * mycophenolate mofetil (MMF), calcineurin inhibitors (CNI) or azathioprine treated patients are eligible if proteinuria is not improving or if kidney function is declining despite treatment with these medications. Once therapy with daratumumab started, these medications need to be discontinued unless they are used as immunosuppressive medication due to renal transplantation.
7. In patients who previously received rituximab, reconstitution of B cells (CD19 normalized, Ly-B-CD19 lab.code 8329) required.
8. Inability to use daratumumab and to comply with the study protocol as assessed by treating nephrologist and/or hematologist (e.g. severe psychiatric illness, severe lung disease, known allergy to daratumumab)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Rate of complete renal remission or partial renal remission and proteinuria and eGFR at EOT. | Through study completion, an average of 12 to 18 months
  Complete renal remission (proteinuria <500 mg/d and <15% decline in baseline eGFR) Partial renal remission (>50% reduction in 24-h proteinuria and < 30% decline in eGFR)

SECONDARY OUTCOMES:
Rate of complete renal remission or partial renal remission and proteinuria and eGFR after 6 cycles of daratumumab. | At the end of daratumumab treatment cycle 6 (each cycle is 28 days)
  Complete renal remission (proteinuria <500 mg/d and <15% decline in baseline eGFR) Partial renal remission (>50% reduction in 24-h proteinuria and < 30% decline in eGFR)
Rate of negativity of bone marrow minimal residual disease (MRD) after 6 and 12 cycles of daratumumab. | At the end of cycle 6 (each cycle is 28 days) and through study completion, an average of 12 to 18 months
Number of patients with complement dysregulation-mediated renal damage caused by paraprotein. | Through study completion, an average of 12 to 18 months
Number of patients in end-stage renal disease or with eGFR decline > 50 %. | Through study completion, an average of 12 to 18 months
Number of patients with proteinuria decline < 25 %. | Through study completion, an average of 12 to 18 months
Number of patients with complete or partial or very good partial hematological remission | Through study completion, an average of 12 to 18 months
Number of patients with serious adverse events (SAE) | Through study completion, an average of 12 to 18 months
Number of patients with significant adverse events (AE) | Through study completion, an average of 12 to 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided